CLINICAL TRIAL: NCT03321422
Title: Lateral Shelf Acetabuloplasty for Treatment of Older Children With Perthes Disease
Brief Title: Lateral Shelf Acetabuloplasty in Perthes Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hesham Mohamed Elbaseet, principal investigator, Assiut University
Other Study IDs: LSAP
Record Dates: First submitted 2017-10-23; First posted 2017-10-25 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Orthopedic Disorder
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention Observational study — follow up of the function of the hip after lateral shelf acetabuloplasty by harris hip score and WOMAC score

SUMMARY:
The incidence of Legg-Calvé-Perthes disease (LCPD) ranges from 0.4/100,000 to 29.0/100,000 children <15 years of age. There is significant variability in incidence within racial groups and is frequently higher in lower socioeconomic classes. The typical age at presentation ranges from 4 to 8 years (average 6.5 years).The optimal treatment goal in Legg-Calvé-Perthes disease (LCPD) is to obtain a spherical femoral head with good congruency to prevent or delay the onset of osteoarthritis after skeletal maturity. There is agreement that patients younger than 5years with a good remodeling capacity have a particularly excellent prognosis, irrespective of treatment.

DETAILED DESCRIPTION:
Older children more than 8 years usually have a poor prognosis, especially without treatment. Apart from the age at diagnosis and surgery, the severity of femoral head flattening and the signs of "head at risk" are also associated with the final clinical outcome. The current surgical treatment options, including proximal femoral varus osteotomy, innominate osteotomy, lateral shelf acetabuloplasty,triple pelvic osteotomy, and Chiari pelvic osteotomy have proved to be effective in covering the femoral head within the acetabulum. To promote the coverage of the femoral head, shelf acetabuloplasty directly increases the size of the acetabulum by implanting graft bone to the lateral rim. When used as salvage surgery, it may provide relief from pain and benefit the involved hip via femoral head flattening, especially in older children. It also improves the spherical remodeling of the femoral head and acetabulum by stimulating lateral acetabular growth. Lateral shelf acetabuloplasty is able to increase the coverage of the femoral head, which is an important tissue for remodeling and preventing further femoral head deformation.

ELIGIBILITY:
Inclusion Criteria:

* Age between 8 up to 14 years
* Patients with Perthes disease and hinged abduction .
* Written consent, free and informed

Exclusion Criteria:

* Age below 8 or above 14 years
* Patients without hinged abduction based on clinical exam and arthrogram under general anaesthesia
* Epiphyseal dysplasia
* Coagulopathy
* Unfit for surgery

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All patients will be admitted at orthopedic department of assiut university hospital. Clinical examination of the hip will be applied. Preoperative hip x ray anteroposterior and lateral views, Radiological classification and grading and clinical evaluation by Harris hip score.
  Hip arthrogram under general anasthesia . if hinged abduction shelf acetabuloplasty will be done. Follow up by x ray and harris hip score at regular visits ( 1.5, 6, 12,24 months)
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Harris hip score | 6 months
  Harris hip score is one of the most commonly used hip score for assessment of hip function.It assess the following items:Pain,support,distance walked, limp, activities-shoes and socks,stairs, public transportation, sitting,flexion deformity, abduction, adduction and external rotation range.The score of these items are summed together to get the total score. Grading according to this score as follows:
  <70= Poor ,70 - 79= Fair, 80-89=Good, 90 -100=Excellent.

CONTACTS AND LOCATIONS:
Locations (1):
- AssiutU, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chaudhry S, Phillips D, Feldman D. Legg-Calve-Perthes disease: an overview with recent literature. Bull Hosp Jt Dis (2013). 2014;72(1):18-27. PMID 25150324
- [Background] Li WC, Xu RJ. Lateral shelf acetabuloplasty for severe Legg-Calve-Perthes disease in patients older than 8 years: A mean eleven-year follow-up. Medicine (Baltimore). 2016 Nov;95(45):e5272. doi: 10.1097/MD.0000000000005272. PMID 27828848
- [Background] Jacobs R, Moens P, Fabry G. Lateral shelf acetabuloplasty in the early stage of Legg-Calve-Perthes disease with special emphasis on the remaining growth of the acetabulum: a preliminary report. J Pediatr Orthop B. 2004 Jan;13(1):21-8. doi: 10.1097/00009957-200401000-00004. PMID 15091254